CLINICAL TRIAL: NCT00970697
Title: Double Blind Randomized Controlled Trial of Recombinant Human Platelet Derived Growth Factor-BB Gel (Regranex Gel®) Versus Hydrogel (Duoderm Hydrogel®) for Healing of MARTORELL's Hypertensive Leg Ulcers. ERAN Trial.
Brief Title: Becaplermin Gel for MARTORELL's Hypertensive Leg Ulcers
Acronym: ERAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P020706
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-09

CONDITIONS: MARTORELL'S ULCER; Hypertensive Leg Ulcer; Necrotic Angiodermatitis
Keywords: MARTORELL'S ULCER; hydrogel; Hypertensive leg ulcer
MeSH Terms: interventions — Bandages, Hydrocolloid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- becaplermin gel (Experimental): application of a continuous thin layer of becaplermin gel (Regranex Gel®) during 8 weeks. The amount of the gel to be applied was determined based on ulcer area at inclusion, and remains identical during all the treatment.
  Interventions: Drug: becaplermin gel
- Duoderm Hydrogel™ (Active Comparator): application of a continuous thin layer of hydrogel dressing (Duoderm Hydrogel®), during 8 weeks. Duoderm Hydrogel™ is a sodium carboxymethylcellulose aqueous-based gel, similar in composition to becaplermin excipient.
  Interventions: Drug: Duoderm Hydrogel™

INTERVENTIONS:
Drug: becaplermin gel — the amount of the gel to be applied was determined based on ulcer area at inclusion and remains identical during all the treatment The posology was identical to what is recommended for Regranex gel®: a single 15g-tube is enough to treat a 5 cm2-wound during 6 weeks (1 cm of gel is applied daily for 5 cm2) Wound was then recovered by a moist saline gauze and a bandage. Becaplermin gel is packaged into masked 15g-tubes.
  Arms: becaplermin gel
Drug: Duoderm Hydrogel™ — The amount of the gel to be applied was determined based on ulcer area at inclusion, and remains identical during all the treatment. The posology was identical to what is recommended for Regranex gel®: a single 15g-tube is enough to treat a 5 cm2-wound during 6 weeks (1 cm of gel is applied daily for 5 cm2) Wound was then recovered by a moist saline gauze and a bandage. Hydrogel dressing is identical in appearance, color, consistency, and odor than becaplermin gel, and packaged in similar masked15g-tubes.
  Arms: Duoderm Hydrogel™

SUMMARY:
Background: No medical treatment has proved its efficacy for the treatment of hypertensive leg ulcers in a well designed trial.

Primary aim of the study: to compare the rate of healing in hypertensive leg ulcers treated with becaplermin gel (Regranex Gel®) daily application versus the application of the same quantity of an hydrogel (Duoderm Hydrogel™), corresponding to the excipient of becaplermin gel.

Method: Ambulatory or hospitalized patients presenting with an hypertensive leg ulcer, were randomized to receive either a daily application of becaplermin gel or hydrogel during 8 weeks. At week 8, a pinch graft was proposed to patients whom the ulcer has not healed.

Primary aim of the study: Complete closure at week 8

Secondary aims: percentage of wound area reduction at week 8, complete closure at week 12, pain and quality of life during treatment

Study hypothesis: becaplermin gel may promote the healing of hypertensive leg ulcers and be an alternative medical treatment to the skin graft usually proposed

DETAILED DESCRIPTION:
Hypertensive leg ulcers are a variety of leg ulcer characterized by very painful and spreading lesions, related to cutaneous microangiopathy, occurring in patients presenting hypertension and /or diabetes. Healing takes a mean of 4 to 12 months. Current treatment is difficult and usually surgical (pinch or meshed skin grafts). Growth factors release by autografted skin may be a significant factor in the promotion of hypertensive leg ulcer healing. Recombinant human platelet derived growth-factor-BB gel (becaplermin gel) has been shown to be effective in the treatment of diabetic ulcers related to diabetic microangiopathy. The objective of the study was to assess the efficacy of becaplermin gel for the healing of hypertensive leg ulcers. Study design: prospective, randomized, multi-centre, double blind, controlled, parallel groupPrimary aim: complete wound closure at week 8Secondary aims: complete wound closure at week 12, pain and quality of life assessment during the treatment( W4,8,10,12), % of wound area reduction at week 8 and 12 Method: Inclusion of 64 patients, 32 in each group. The study population consisted of consecutive patients presenting with one or more leg ulcers diagnosed as hypertensive MARTORELL's ulcers: hypertensive and/or diabetic patients, in absence of chronic venous insufficiency (C5-C6 of the CEAP) or peripheral arterial occlusive disease (presence of peripheral pulses or ankle brachial index ≥0.8), superficial spreading necrotic ulcer, presence of spontaneous pain, and presence of a red purpuric margin. Treatment consists of a daily application of a continuous thin layer of becaplermin gel (Regranex Gel®) or Duoderm Hydrogel™, during 8 weeks. The amount of the gel to be applied was determined based on ulcer area at inclusion (as recommended for Regranex gel®), and remains identical during all the treatment. Wound was then recovered by a moist saline gauze and a bandage. Duoderm Hydrogel™ is a sodium carboxymethylcellulose aqueous-based gel, similar in composition to becaplermin excipient.At week 8, a pinch graft was proposed to patients whom the ulcer was not healed. Between weeks 8 and 12, if patient had not healed and was not grafted, dressing was chosen by the investigator, depending on the wound stage. All patients were followed until week 12.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years of age or older, able to give informed consent and to follow the treatment procedure
* target ulcer area between 1 and 30 cm2
* consecutive patients presenting with one or more leg ulcers diagnosed as hypertensive MARTORELL's ulcers
* presence of an arterial hypertension, according to the WHO criteria, treated or not; and/or presence of a diabetes treated by oral agent, insulin or diet
* absence of clinical signs of chronic venous insufficiency: skin hyperpigmentation, lipodermatosclerosis
* absence of significant peripheral arterial occlusive disease: presence of peripheral pulses or ankle brachial index ≥0.8
* absence of clinical sign of arterial insufficiency: intermittent claudication, resting pain
* superficial spreading necrotic ulcer
* presence of spontaneous pain
* presence of a red purpuric margin

Exclusion Criteria:

* pregnancy
* allergy to hydrogel or to becaplermin gel
* uncontrolled or evolving systemic disease: cardiac or renal failure, hepatic insufficiency, malignant disease, thrombotic disease, vasculitis or other connective tissue disorder
* presence of a cryoglobulinemia
* serum creatinine concentration greater than 200µmol/L or uncontrolled diabetes (fasting blood glucose > 2,5 g/L under treatment)
* concomitant treatment by ILOMEDINE
* bone, joint or tendon (except for achilles tendon) exposition in the wound
* systemic treatment with corticosteroid agents or cytotoxic drugs in the past 3 months before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-01; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Complete wound closure rate at week 8 of treatment | week 9

SECONDARY OUTCOMES:
Complete wound closure rate at week 12 of treatment | week 13
pain and quality of life evolution during the treatment( W4,8,10,12), | week 9
% of wound area reduction at week 8 and 12 | weeks 9 and 13
safety of the treatment at week 4, 8 and 12 | week 13

CONTACTS AND LOCATIONS:
Overall Officials: Patricia SENET, Principal Investigator — Dermatology, Charles Foix
Locations (1):
- Hospital Charles Foix, Ivry-sur-Seine, Île-de-France Region, France

REFERENCES:
- [Derived] Senet P, Vicaut E, Beneton N, Debure C, Lok C, Chosidow O. Topical treatment of hypertensive leg ulcers with platelet-derived growth factor-BB: a randomized controlled trial. Arch Dermatol. 2011 Aug;147(8):926-30. doi: 10.1001/archdermatol.2011.84. Epub 2011 Apr 11. PMID 21482863